CLINICAL TRIAL: NCT04445051
Title: Exploratory Investigation on Performance and Safety of New Intermittent Catheters in Healthy Volunteers
Brief Title: Investigation of New Intermittent Catheters in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CP322
Record Dates: First submitted 2020-05-28; First posted 2020-06-24 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2022-08

CONDITIONS: Retention, Urinary
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intermittent catheter; SpeediCath® Standard male or female (Active Comparator): Participants underwent catheterization with standard of care intermittent catheter. The catheterization was performed by a trained nurse.
  Interventions: Device: SpeediCath® Standard male or female
- New intermittent catheter Variant 1 for male or female (Experimental): Participants underwent catheterization with the new intermittent catheter Variant 1 for males or females. The catheterization was performed by a trained nurse.
  Interventions: Device: New intermittent Variant 1 catheter for male or female
- New intermittent catheter Variant 2 for male or female (Experimental): Participants underwent catheterization with the new intermittent catheter Variant 2 for males or females. The catheterization was performed by a trained nurse.
  Interventions: Device: New intermittent Variant 2 catheter for male or female

INTERVENTIONS:
Device: SpeediCath® Standard male or female — Intermittent catheterization through the urethra draining the bladder, using SpeediCath® Standard male or female.
  Arms: Intermittent catheter; SpeediCath® Standard male or female
Device: New intermittent Variant 1 catheter for male or female — Intermittent catheterization through the urethra draining the bladder, using the new Variant 1 for male or female.
  Arms: New intermittent catheter Variant 1 for male or female
Device: New intermittent Variant 2 catheter for male or female — Intermittent catheterization through the urethra draining the bladder, using the new Variant 2 for male or female.
  Arms: New intermittent catheter Variant 2 for male or female

SUMMARY:
Investigation of non-CE marked intermittent catheters. The study was a randomized, single blinded, cross-over investigation comparing two new catheters with a comparator catheter in 30 adult healthy volunteers.

DETAILED DESCRIPTION:
The CP322 study investigated a novel non-CE marked intermittent catheter for males and females, designed in two different variants, Variant 1 and Variant 2, respectively. The study was conducted in Denmark and was a randomized, single blinded, cross-over investigation comparing the two new variant catheters with a comparator catheter in 30 adult healthy volunteers.

For each participant, the study thus contained three test visits/treatment arms (Comparator, Variant 1 and Variant 2, respectively), to which the 30 participants were randomized using a randomization sequence of six (i.e., there were six different random options for the order in which the participants tested the three catheters). There were 4-14 days between the test visits.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years of age and with full legal capacity
* Written informed consent and signed letter of authority and secrecy agreement given
* Willing to comply with not using analgesics 1 up to 24 hours prior to catheterization visits
* Urine Multistix negative for erythrocytes (hematuria)

Exclusion Criteria:

* Participation in any other clinical investigations during this investigation
* Known hypersensitivity towards any of the test products
* Symptoms of urinary tract infection (UTI) (Investigators judgement)
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Bagi, MD, Principal Investigator — Blegdamsvej 9, Urologisk klinik Afsnit 2112, Rigshospitalet, Denmark
Locations (1):
- Urologisk klinik, Afsnit 2112, Rigshospitalet, Copenhagen, Copenhagen Ø, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Landauro MH, Tentor F, Pedersen T, Jacobsen L, Bagi P. Improved Performance With the Micro-Hole Zone Intermittent Catheter: A Combined Analysis of 3 Randomized Controlled Studies Comparing the New Catheter Technology With a Conventional Eyelet Catheter. J Wound Ostomy Continence Nurs. 2023 Nov-Dec 01;50(6):504-511. doi: 10.1097/WON.0000000000001029. PMID 37966080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 2020 and September 2020, 30 users were recruited for the study from one site (Denmark) and encompassed the safety population.
Pre-assignment Details: The 30 recruited participant were randomized into the three treatment arms, using a randomization sequence of six. No participants were excluded, one was discontinued after Visit 2 due to an adverse event.
  Two participants total had an adverse event, both were classified as mild, non-serious, 'Possibly related' and 'Not related' (for details; see Adverse Events section).
  Thus, 30 participants constituted the intention to treat (ITT) population.
Groups:
- Comparator, Then Variant 2, Then Variant 1: On three separate visits and in the listed random order, the participants underwent three interventions:
  First intervention: Day of catheterization with Comparator. Washout: 4-14 days. Second intervention: Day of catheterization with Variant 2. Washout: 4-14 days. Third intervention: Day of catheterization with Variant 1.
- Variant 2, Then Variant 1, Then Comparator: On three separate visits and in the listed random order, the participants underwent three interventions:
  First intervention: Day of catheterization with Variant 2. Washout: 4-14 days. Second intervention: Day of catheterization with Variant 1. Washout: 4-14 days. Third intervention: Day of catheterization with Comparator.
- Comparator, Then Variant 1, Then Variant 2: On three separate visits and in the listed random order, the participants underwent three interventions:
  First intervention: Day of catheterization with Comparator. Washout: 4-14 days. Second intervention: Day of catheterization with Variant 1. Washout: 4-14 days. Third intervention: Day of catheterization with Variant 2.
- Variant 1, Then Comparator, Then Variant 2: On three separate visits and in the listed random order, the participants underwent three interventions:
  First intervention: Day of catheterization with Variant 1. Washout: 4-14 days. Second intervention: Day of catheterization with Comparator. Washout: 4-14 days. Third intervention: Day of catheterization with Variant 2.
- Variant 1, Then Variant 2, Then Comparator: On three separate visits and in the listed random order, the participants underwent three interventions:
  First intervention: Day of catheterization with Variant 1. Washout: 4-14 days. Second intervention: Day of catheterization with Variant 2. Washout: 4-14 days. Third intervention: Day of catheterization with Comparator.
- Variant 2, Then Comparator, Then Variant 1: On three separate visits and in the listed random order, the participants underwent three interventions:
  First intervention: Day of catheterization with Variant 2. Washout: 4-14 days. Second intervention: Day of catheterization with Comparator. Washout: 4-14 days. Third intervention: Day of catheterization with Variant 1.
Period: Overall Study
Arm/Group | Comparator, Then Variant 2, Then Variant 1 | Variant 2, Then Variant 1, Then Comparator | Comparator, Then Variant 1, Then Variant 2 | Variant 1, Then Comparator, Then Variant 2 | Variant 1, Then Variant 2, Then Comparator | Variant 2, Then Comparator, Then Variant 1
Started | 5 | 4 | 5 | 6 | 5 | 5
Completed | 5 | 4 | 4 | 6 | 5 | 5
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Female ITT Population: Each treatment arm consisted of three test visits with 4-14 days between each crossover. On each visit, the participants underwent intermittent catheterization through the urethra, draining the bladder, and tested a different intermittent catheter: The comparator catheter (SpeediCath® Standard female), the new Variant 1 female catheter, or the new Variant 2 female catheter.
- Male ITT Population: Each treatment arm consisted of three test visits with 4-14 days between each crossover. On each visit, the participants underwent intermittent catheterization through the urethra, draining the bladder, and tested a different intermittent catheter: The comparator catheter (SpeediCath® Standard male), the new Variant 1 male catheter, or the new Variant 2 male catheter.
- Total: Total of all reporting groups
Arm/Group | Female ITT Population | Male ITT Population | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (12) | 32 (8) | 32 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 0 | 15
  Male | 0 | 15 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 15 | 15 | 30
Hematuria positive [Count of Participants; unit: Participants] — Blood in the urine; dipstick analysis positive.
  Participants | 0 | 0 | 0
Hematuria negative [Count of Participants; unit: Participants] — Blood in the urine; dipstick analysis negative.
  Participants | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Residual Urine at 1st Flow-stop
Description: The residual urine at 1st flow-stop during catheterization (performed by a nurse) represents the volume of urine left in the bladder, the first time the urine stops running out of the catheter during bladder emptying/urination. This was assessed using a pressure sensor with time-logged weighing, meaning that a flow-stop was registered measuring the hydrostatic pressure at the outlet of an intermittent urinary catheter. Simultaneously, the collected urine was weighed and converted to volume, and the residual volume at first flow stop was calculated as the difference between the total urine volume collected and the volume collected at the first flow-stop.
Time Frame: Immediately after the procedure/catheterization, up to 5 min.
Population: The intention to treat population (full analysis set) constituted all randomized subjects with a valid informed consent who was exposed to at least one product, and with valid information on at least one product with respect to the endpoints.
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Intermittent Catheter; SpeediCath® Standard Female: Female participants underwent intermittent catheterization through the urethra, draining the bladder. Catheterization was performed with standard of care intermittent catheter; SpeediCath® Standard female (active comparator). The catheterizations were performed by a trained nurses.
- New Intermittent Catheter Variant 1 for Female: Female participants underwent intermittent catheterization through the urethra, draining the bladder. Catheterization was performed with new intermittent catheter Variant 1 for females. The catheterizations were performed by a trained nurses.
- New Intermittent Catheter Variant 2 for Female: Female participants underwent intermittent catheterization through the urethra, draining the bladder. Catheterization was performed with new intermittent catheter Variant 2 for females. The catheterizations were performed by a trained nurses.
- Intermittent Catheter; SpeediCath® Standard Male: Male participants underwent intermittent catheterization through the urethra, draining the bladder. Catheterization was performed with standard of care intermittent catheter; SpeediCath® Standard male (active comparator). The catheterizations were performed by a trained nurses.
- New Intermittent Catheter Variant 1 for Male: Male participants underwent intermittent catheterization through the urethra, draining the bladder. Catheterization was performed with new intermittent catheter Variant 1 for males. The catheterizations were performed by a trained nurses.
- New Intermittent Catheter Variant 2 for Male: Male participants underwent intermittent catheterization through the urethra, draining the bladder. Catheterization was performed with new intermittent catheter Variant 2 for males. The catheterizations were performed by a trained nurses.
Arm/Group | Intermittent Catheter; SpeediCath® Standard Female | New Intermittent Catheter Variant 1 for Female | New Intermittent Catheter Variant 2 for Female | Intermittent Catheter; SpeediCath® Standard Male | New Intermittent Catheter Variant 1 for Male | New Intermittent Catheter Variant 2 for Male
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
mL | 35.0 (71.0) | 1.1 (2.6) | 0.2 (0.7) | 37.0 (40.0) | 2.2 (6.2) | 1.0 (4.0)
Statistical Analysis 1: Comparison: Intermittent Catheter; SpeediCath® Standard Female vs New Intermittent Catheter Variant 1 for Female; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.010, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; Random effect: Subject. Fixed effects: Visit (Visit 1, 2 and 3), Treatment (comparator, Variant 1 and Variant 2)*Gender (male and females); Mean Difference (Final Values) = 32.9, 95% CI 2-sided [8.3 to 57.5]
Statistical Analysis 2: Comparison: Intermittent Catheter; SpeediCath® Standard Female vs New Intermittent Catheter Variant 2 for Female; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.007, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 34.3, 95% CI 2-sided [9.8 to 58.8]
Statistical Analysis 3: Comparison: New Intermittent Catheter Variant 1 for Female vs New Intermittent Catheter Variant 2 for Female; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.908, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-23.1 to 25.9]
Statistical Analysis 4: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 1 for Male; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.006, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 35.3, 95% CI 2-sided [10.8 to 59.8]
Statistical Analysis 5: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 2 for Male; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.005, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 36.8, 95% CI 2-sided [11.9 to 61.8]
Statistical Analysis 6: Comparison: New Intermittent Catheter Variant 1 for Male vs New Intermittent Catheter Variant 2 for Male; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.899, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-23.3 to 26.5]

2. Secondary Outcome: Post-void Residual Urine
Description: The volume of residual urine (urine left in the bladder) post catheterization (performed by the nurse) measured in triplicates using an ultrasound scanner.
Time Frame: Immediately after the procedure/catheterization, up to 15 min.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Intermittent Catheter; SpeediCath® Standard Female | New Intermittent Catheter Variant 1 for Female | New Intermittent Catheter Variant 2 for Female | Intermittent Catheter; SpeediCath® Standard Male | New Intermittent Catheter Variant 1 for Male | New Intermittent Catheter Variant 2 for Male
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
mL | 8.6 (11.4) | 1.5 (6.1) | 27.6 (104.1) | 5.3 (8.9) | 24.3 (79.1) | 16.3 (31.9)
Statistical Analysis 1: Comparison: Intermittent Catheter; SpeediCath® Standard Female vs New Intermittent Catheter Variant 1 for Female; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.665, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 8.8, 95% CI 2-sided [-31.9 to 49.6]
Statistical Analysis 2: Comparison: Intermittent Catheter; SpeediCath® Standard Female vs New Intermittent Catheter Variant 2 for Female; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.375, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -18.1, 95% CI 2-sided [-58.7 to 22.4]
Statistical Analysis 3: Comparison: New Intermittent Catheter Variant 1 for Female vs New Intermittent Catheter Variant 2 for Female; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.188, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -27.0, 95% CI 2-sided [-67.6 to 13.6]
Statistical Analysis 4: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 1 for Male; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.361, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -18.6, 95% CI 2-sided [-59.3 to 21.9]
Statistical Analysis 5: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 2 for Male; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.600, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -10.9, 95% CI 2-sided [-52.3 to 30.5]
Statistical Analysis 6: Comparison: New Intermittent Catheter Variant 1 for Male vs New Intermittent Catheter Variant 2 for Male; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.707, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 7.78, 95% CI 2-sided [-33.5 to 49.0]

3. Secondary Outcome: Catheterization Insertion Discomfort
Description: Discomfort measured at catheter insertion, using the Visual Analogue Scale (VAS). The VAS is a tool used to rate the intensity of certain sensations and feelings, e.g. discomfort/pain. It is a straight line of 10 cm (in this case horizontal) with one end meaning no discomfort/pain (0 cm) and the other end meaning the worst discomfort/pain imaginable (10 cm). The subject visualizes and marks a point on the line that matches the amount of discomfort/pain experienced. A high score reflects a worse outcome than a lower score.
Time Frame: Immediately after the procedure/catheterization, up to 5 min.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intermittent Catheter; SpeediCath® Standard Female | New Intermittent Catheter Variant 1 for Female | New Intermittent Catheter Variant 2 for Female | Intermittent Catheter; SpeediCath® Standard Male | New Intermittent Catheter Variant 1 for Male | New Intermittent Catheter Variant 2 for Male
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
cm | 0.51 (0.72) | 0.81 (0.96) | 0.86 (1.15) | 2.32 (2.24) | 2.31 (1.97) | 2.79 (2.46)
Statistical Analysis 1: Comparison: Intermittent Catheter; SpeediCath® Standard Female vs New Intermittent Catheter Variant 1 for Female; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.615, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-1.08 to 0.65]
Statistical Analysis 2: Comparison: Intermittent Catheter; SpeediCath® Standard Female vs New Intermittent Catheter Variant 2 for Female; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.480, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-1.17 to 0.56]
Statistical Analysis 3: Comparison: New Intermittent Catheter Variant 1 for Female vs New Intermittent Catheter Variant 2 for Female; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.839, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.95 to 0.77]
Statistical Analysis 4: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 1 for Male; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.894, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.92 to 0.80]
Statistical Analysis 5: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 2 for Male; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.195, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-1.46 to 0.30]
Statistical Analysis 6: Comparison: New Intermittent Catheter Variant 1 for Male vs New Intermittent Catheter Variant 2 for Male; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.242, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-1.40 to 0.36]

4. Secondary Outcome: Catheterization Urination Discomfort
Description: Discomfort measured during catheter emptying/urination, using the Visual Analogue Scale (VAS). The VAS is a tool used to rate the intensity of certain sensations and feelings, e.g. discomfort/pain. It is a straight line of 10 cm (in this case horizontal) with one end meaning no discomfort/pain (0 cm) and the other end meaning the worst discomfort/pain imaginable (10 cm). The subject visualizes and marks a point on the line that matches the amount of discomfort/pain experienced. A high score reflects a worse outcome than a lower score.
Time Frame: Immediately after the procedure/catheterization, up to 5 min.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intermittent Catheter; SpeediCath® Standard Female | New Intermittent Catheter Variant 1 for Female | New Intermittent Catheter Variant 2 for Female | Intermittent Catheter; SpeediCath® Standard Male | New Intermittent Catheter Variant 1 for Male | New Intermittent Catheter Variant 2 for Male
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
cm | 0.18 (0.23) | 0.47 (0.83) | 0.55 (0.93) | 0.93 (1.62) | 0.74 (0.86) | 1.51 (2.77)
Statistical Analysis 1: Comparison: Intermittent Catheter; SpeediCath® Standard Female vs New Intermittent Catheter Variant 1 for Female; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.639, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-1.20 to 0.74]
Statistical Analysis 2: Comparison: Intermittent Catheter; SpeediCath® Standard Female vs New Intermittent Catheter Variant 2 for Female; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.492, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-1.30 to 0.63]
Statistical Analysis 3: Comparison: New Intermittent Catheter Variant 1 for Female vs New Intermittent Catheter Variant 2 for Female; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.828, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-1.07 to 0.86]
Statistical Analysis 4: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 1 for Male; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.744, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.81 to 1.13]
Statistical Analysis 5: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 2 for Male; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.208, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-1.62 to 0.36]
Statistical Analysis 6: Comparison: New Intermittent Catheter Variant 1 for Male vs New Intermittent Catheter Variant 2 for Male; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.116, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.79, 95% CI 2-sided [-1.77 to 0.20]

5. Secondary Outcome: Withdrawal Discomfort
Description: Discomfort measured during catheter withdrawal, using the Visual Analogue Scale (VAS). The VAS is a tool used to rate the intensity of certain sensations and feelings, e.g. discomfort/pain. It is a straight line of 10 cm (in this case horizontal) with one end meaning no discomfort/pain (0 cm) and the other end meaning the worst discomfort/pain imaginable (10 cm). The subject visualizes and marks a point on the line that matches the amount of discomfort/pain experienced. A high score reflects a worse outcome than a lower score.
Time Frame: Immediately after the procedure/catheterization, up to 5 min.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intermittent Catheter; SpeediCath® Standard Female | New Intermittent Catheter Variant 1 for Female | New Intermittent Catheter Variant 2 for Female | Intermittent Catheter; SpeediCath® Standard Male | New Intermittent Catheter Variant 1 for Male | New Intermittent Catheter Variant 2 for Male
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
cm | 0.79 (0.70) | 0.83 (0.94) | 1.11 (1.32) | 2.05 (2.55) | 1.42 (1.86) | 2.28 (2.39)
Statistical Analysis 1: Comparison: Intermittent Catheter; SpeediCath® Standard Female vs New Intermittent Catheter Variant 1 for Female; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.798, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.75 to 0.96]
Statistical Analysis 2: Comparison: Intermittent Catheter; SpeediCath® Standard Female vs New Intermittent Catheter Variant 2 for Female; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.556, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-1.10 to 0.60]
Statistical Analysis 3: Comparison: New Intermittent Catheter Variant 1 for Female vs New Intermittent Catheter Variant 2 for Female; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.399, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-1.21 to 0.49]
Statistical Analysis 4: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 1 for Male; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.198, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.55, 95% CI 2-sided [-0.30 to 1.41]
Statistical Analysis 5: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 2 for Male; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.365, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-1.27 to 0.48]
Statistical Analysis 6: Comparison: New Intermittent Catheter Variant 1 for Male vs New Intermittent Catheter Variant 2 for Male; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.033, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.95, 95% CI 2-sided [-1.82 to -0.08]

6. Secondary Outcome: Overall Catheterization Discomfort
Description: Discomfort measured for the overall/entire catheterization procedure, using the Visual Analogue Scale (VAS). The VAS is a tool used to rate the intensity of certain sensations and feelings, e.g. discomfort/pain. It is a straight line of 10 cm (in this case horizontal) with one end meaning no discomfort/pain (0 cm) and the other end meaning the worst discomfort/pain imaginable (10 cm). The subject visualizes and marks a point on the line that matches the amount of discomfort/pain experienced. A high score reflects a worse outcome than a lower score.
Time Frame: Immediately after the procedure/catheterization, up to 5 min.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intermittent Catheter; SpeediCath® Standard Female | New Intermittent Catheter Variant 1 for Female | New Intermittent Catheter Variant 2 for Female | Intermittent Catheter; SpeediCath® Standard Male | New Intermittent Catheter Variant 1 for Male | New Intermittent Catheter Variant 2 for Male
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
cm | 0.66 (0.65) | 0.72 (0.63) | 1.04 (1.63) | 1.99 (2.19) | 1.71 (1.57) | 2.58 (2.56)
Statistical Analysis 1: Comparison: Intermittent Catheter; SpeediCath® Standard Female vs New Intermittent Catheter Variant 1 for Female; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.882, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.83 to 0.96]
Statistical Analysis 2: Comparison: Intermittent Catheter; SpeediCath® Standard Female vs New Intermittent Catheter Variant 2 for Female; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.478, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-1.21 to 0.57]
Statistical Analysis 3: Comparison: New Intermittent Catheter Variant 1 for Female vs New Intermittent Catheter Variant 2 for Female; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.391, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-1.27 to 0.51]
Statistical Analysis 4: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 1 for Male; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.657, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.69 to 1.09]
Statistical Analysis 5: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 2 for Male; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.125, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-1.62 to 0.20]
Statistical Analysis 6: Comparison: New Intermittent Catheter Variant 1 for Male vs New Intermittent Catheter Variant 2 for Male; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.051, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.91, 95% CI 2-sided [-1.81 to 0.00]

7. Secondary Outcome: Post-catheterization Urination Discomfort
Description: Discomfort measured for the first normal void/urination after the catheterization procedure, using the Visual Analogue Scale (VAS). The VAS is a tool used to rate the intensity of certain sensations and feelings, e.g. discomfort/pain. It is a straight line of 10 cm (in this case horizontal) with one end meaning no discomfort/pain (0 cm) and the other end meaning the worst discomfort/pain imaginable (10 cm). The subject visualizes and marks a point on the line that matches the amount of discomfort/pain experienced. A high score reflects a worse outcome than a lower score.
Time Frame: Immediately after the first normal void following the procedure/catheterization, up to 5 min.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intermittent Catheter; SpeediCath® Standard Female | New Intermittent Catheter Variant 1 for Female | New Intermittent Catheter Variant 2 for Female | Intermittent Catheter; SpeediCath® Standard Male | New Intermittent Catheter Variant 1 for Male | New Intermittent Catheter Variant 2 for Male
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
cm | 0.29 (0.63) | 0.09 (0.16) | 0.35 (0.72) | 0.66 (1.56) | 0.66 (0.84) | 1.88 (2.70)
Statistical Analysis 1: Comparison: Intermittent Catheter; SpeediCath® Standard Female vs New Intermittent Catheter Variant 1 for Female; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.877, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.83 to 0.97]
Statistical Analysis 2: Comparison: Intermittent Catheter; SpeediCath® Standard Female vs New Intermittent Catheter Variant 2 for Female; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.351, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-1.31 to 0.47]
Statistical Analysis 3: Comparison: New Intermittent Catheter Variant 1 for Female vs New Intermittent Catheter Variant 2 for Female; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.278, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-1.38 to 0.40]
Statistical Analysis 4: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 1 for Male; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.711, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.73 to 1.06]
Statistical Analysis 5: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 2 for Male; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.024, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.06, 95% CI 2-sided [-1.97 to -0.15]
Statistical Analysis 6: Comparison: New Intermittent Catheter Variant 1 for Male vs New Intermittent Catheter Variant 2 for Male; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.009, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.23, 95% CI 2-sided [-2.14 to -0.31]

ADVERSE EVENTS:
Time Frame: Each participant was enrolled for 3 x 4-14 days for the entire investigation, thus a maximum of 42 days.
Description: The relationship to the investigational or comparator products was collected. The safety population constituted the subjects who had given informed consent and were thus 30 participants.
  An adverse event was reported as either: "Not related", "Unlikely related", "Possibly related", "Probably related", or "Definitely related", to the comparator to the Variant 1 or Variant 2 products.
Arm/Group | Intermittent Catheter; SpeediCath® Standard Female | New Intermittent Catheter Variant 1 for Female | New Intermittent Catheter Variant 2 for Female | Intermittent Catheter; SpeediCath® Standard Male | New Intermittent Catheter Variant 1 for Male | New Intermittent Catheter Variant 2 for Male
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 1/15 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intermittent Catheter; SpeediCath® Standard Female (N=15) | New Intermittent Catheter Variant 1 for Female (N=15) | New Intermittent Catheter Variant 2 for Female (N=15) | Intermittent Catheter; SpeediCath® Standard Male (N=15) | New Intermittent Catheter Variant 1 for Male (N=15) | New Intermittent Catheter Variant 2 for Male (N=14)
Possibly related (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Urinary tract infection (UTI)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT04445051/Prot_SAP_000.pdf